CLINICAL TRIAL: NCT05532826
Title: Clinical Study on the Efficacy and Safety of Donor EBV-CTL Infusion in Patients With CAEBV and EBV-associated Hemophagocytic Lymphohistiocytosis After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Clinical Study of Donor EBV-CTL Infusion in Patients With CAEBV and EBV-HLH After Allo-HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBV-CTL，CAEBV/EBV-HLH
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-09

CONDITIONS: Chronic Active Epstein-Barr Virus Infection; Virus-Associated Hemophagocytic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBV-CTL infusion patients (Experimental): Given donor EBV-CTL infusion after allo HSCT
  Interventions: Other: donor EBV-specific T lymphocytes

INTERVENTIONS:
Other: donor EBV-specific T lymphocytes — EBV-DNA reactive after transplantation, or did not turn negative after +30 days, peripheral blood lymphocytes of the donor were collected to prepare EBV-CTL, and the first transfusion of EBV-CTL 6.0x105 was given at 48h to rapidly culture EBV-CTL, then EBV-CTL 6.0x105/kg was injected once a week untile EBV-DNA negative for 2 consecutive times or GVHD happened. After the second infusion, EBV-DNA did not decrease and there was no aGVHD patients, EBV-CTL infusion volume was increased to 1.2x106/kg, once a week. After 2 cycle infusion, EBV-DNA still did not decrease, and the reinfusion was terminated.
  Peripheral blood lymphocytes were collected from donors of high-risk patients at +14 days after allogeneic hematopoietic stem cell transplantation to prepare EBV-CTL, and EBV-CTL 6.0x105/kg was infused at +21d, +28d, +35d and + 42D for prevention. During treatment, if the patient develops GVHD, the infusion should be stopped.

SUMMARY:
To evaluate the efficacy and safety of donor EBV-specific T lymphocytes (EBV-CTL) infusion in patients with chronic active Epstein-Barr virus infection (CAEBV) and EBV-associated hemophagocytic lymphohistiocytosis (EBV-HLH) after allogeneic hematopoietic stem cell transplantation (allo-HSCT)

DETAILED DESCRIPTION:
Evaluate the efficacy and safety of donor EBV-specific T lymphocytes (EBV-CTL) infusion in patients with chronic active Epstein-Barr virus infection (CAEBV) and EBV-associated hemophagocytic lymphohistiocytosis (EBV-HLH) after allogeneic hematopoietic stem cell transplantation (allo-HSCT)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CAEBV or EBV-HLH who were eligible for allogeneic hematopoietic stem cell transplantation agreed to regular monitoring of EBV-DNA after transplantation.
2. Age ≤65 years old, ECOG score 0-2.
3. Organ function: Cardiac EF≥40%, creatinine clearance ≥50%, aminotransferase (ALT/AST) < 200U/L.
4. The estimated survival time is more than 3 months. 5) Have donors who meet the requirements of allogeneic hematopoietic stem cell transplantation donors， and the donor agreed to collect lymphocytes to prepare EBV-CTL

Exclusion Criteria:

1. The patient or donor had a New York Heart Association (NYHA) score of grade II or higher (including grade II). Or a definite diagnosis of cirrhosis.
2. There are active infections other than EBV that have not yet been controlled.
3. The donor has a blood-borne infectious disease (e.g. HIV, hepatitis B, hepatitis C, syphilis, etc.). The patient was positive for HBV-DNA or HCV-RNA.
4. Active major hemorrhage of internal organs (including gastrointestinal hemorrhage, alveolar hemorrhage, intracranial hemorrhage, etc.).
5. The donor refused to collect lymphocytes to prepare EBV-CTL cells, or the number of EBV-CTL cells prepared from the donor did not meet the infusion requirements.
6. At the same time participate in other clinical studies.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA | 1 year
  EBV-DNA negative conversion rate for patients with relapse/non-remission and EBV-DNA reactivation rate for high-risk patients

CONTACTS AND LOCATIONS:
Overall Officials: zhao wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Zhao Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No